CLINICAL TRIAL: NCT00492388
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study Comparing the Efficacy and Safety of PMI-150 (Intranasal Ketamine) to Placebo as an Analgesic for the Treatment of Breakthrough Pain in Cancer Patients
Brief Title: Safety and Efficacy of PMI-150 (Intranasal Ketamine) for the Treatment of Breakthrough Pain in Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision not to continue development
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-016
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Pain; Cancer
Keywords: breakthrough; pain; cancer
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): PMI-150 (intranasal ketamine)
  Interventions: Drug: PMI-150 (intranasal ketamine)
- B (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PMI-150 (intranasal ketamine) — intranasal dosing
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
To assess the safety and efficacy of PMI-150 (Intranasal Ketamine) as an analgesic for the treatment of breakthrough pain in cancer patients.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and efficacy following the administration of intranasal ketamine in providing pain relief as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* Patients requiring around-the-clock opioids for pain due to cancer and with a history of experiencing episodes of breakthrough pain

Exclusion Criteria:

* under 18 years
* non-cancer pain
* allergy to ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
pain intensity difference | 60 minutes

SECONDARY OUTCOMES:
various pain assessments | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Bajwa, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States